CLINICAL TRIAL: NCT06187701
Title: Pilot Study on the Use of the Co-Active Therapeutic Theatre (Co-ATT) Manualised Model of Drama Therapy for the Treatment of Patients With Co-occurring Primary Psychiatric and Substance Use Disorders
Brief Title: Co-Active Therapeutic Theatre (Co-ATT) for Dual-Diagnosis Patients
Acronym: Co-ATT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43656
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Issue; Substance Use Disorders
Keywords: Drama therapy; Psychiatric symptom severity; Subjective quality of life; Overall functioning
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Co-Active Therapeutic Theatre (Co-ATT) (Experimental): Drama therapy will be used to treat participants with co-occurring primary psychiatric and substance use disorders
  Interventions: Behavioral: Co-Active Therapeutic Theatre (Co-ATT)

INTERVENTIONS:
Behavioral: Co-Active Therapeutic Theatre (Co-ATT) — There will be one group drama therapy session per week, for a total of twelve weeks (i.e., total twelve sessions) followed by a single performance (with composition of the audience determined by unanimous agreement of the participants) of the dramatic work (script) produced by the participants during the course of the drama therapy intervention.

SUMMARY:
Drama Therapy involves of the use of theatrical techniques (such as script development, acting exercises, improvisation, etc.) to help treat patients' mental illness and improve their functioning and overall sense of wellbeing.

This study will evaluate the effectiveness of a specific version of drama therapy for the treatment of patients suffering from both mental illness (such as depression, bipolar disorder, schizophrenia, etc.) and one or more substance use disorders. The study will also assess participants feelings and thoughts about the drama therapy intervention (such as whether or not they enjoyed it and if/how they found it helpful).

The drama therapy intervention will consist of one group drama therapy session per week, for a total of twelve weeks (i.e., total twelve sessions) followed by a single performance (with composition of the audience determined by unanimous agreement of the participants) of the dramatic work (script) produced by the participants during the course of the drama therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with at least one primary psychiatric disorder, and
* Diagnosed with at least one substance use disorder
* Both disorders active (i.e., meeting DSM-V criteria for each disorder (i.e., with ongoing psychiatric symptoms and ongoing substance use)
* Enrolled in the Addiction Psychiatry Treatment Program (APTP) at Boston Medical Center (i.e., scheduled for follow-up appointments with therapist and/or psychiatrist in APTP).
* Currently taking medications and those not currently taking medications

Exclusion Criteria:

* Incarcerated persons
* Pregnant women
* Inability to understand and/or sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in substance use | baseline, 12 weeks
  Assessed with the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool. TAPS consists of a combined screening component (TAPS-1) followed by a brief followed by a brief assessment (TAPS-2) for those who screen positive. Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance. TAPS Score Risk Category- 0=No Use in Past 3 Months, 1=Problem Use, 2+ =Higher Risk
Change in psychiatric symptom severity for a history of Major Depressive Disorder (MDD) | baseline, 12 weeks
  The Patient Health Questionnaire (PHQ) will be used to assess this outcome. It is a multiple-choice self-report inventory that is used as a screening and diagnostic tool for mental health disorders of depression, anxiety, alcohol, eating, and somatoform disorders.There are 9 questions with a score from 0=Not al all to 3=Nearly everyday and one additional question about level of difficulty. Scores can range from 1 to 27 and are interpreted as: 1-4 Minimal depression, 5-9 Mild depression, 10-14 Moderate depression, 15-19 Moderately severe depression, and 20-27 Severe depression.
Change in psychiatric symptom severity given a history of bipolar disorder with the BDRS | baseline, 12 weeks
  The Bipolar Depression Rating Scale (BDRS) has 20 questions with responses from 0= Nil to 3= Severe. The maximum score possible is 60. Higher scores indicate greater severity of symptoms.
Change in psychiatric symptom severity given a history of bipolar disorder with the YMRS | baseline, 12 weeks
  The Young Mania Rating Scale (YMRS) has eleven items and is based on the patient's subjective report of his or her clinical condition, and generally limited to the previous 48 hours. Scores can range from 0 to 60 and higher scores are associated with more severe symptoms.
Change in psychiatric symptom severity for a history of post traumatic stress disorder (PTSD) | baseline, 12 weeks
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) will be used to assess this outcome. The total severity score on the CAPS-5 represents the sum of the individual severity scores (0-4) for each of the 20 PTSD symptoms. Total scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Change in psychiatric symptom severity for a history of schizophrenia/schizophrenic disorders. | baseline, 12 weeks
  The Positive and Negative Syndrome Scale (PANSS) will be used to asses this outcome. PANSS items are rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme); because the absence of symptoms is equal to 1 point, the lowest possible total score on both PANSS scales is 7. The range for both the negative and positive scales are 7 to 49.
Change in subjective quality of life | baseline, 12 weeks
  The Quality of Life Scale (QOLS) will be used to assess this outcome. The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112. Higher score indicate higher quality of life.
Change in overall functioning | baseline, 12 weeks
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) will be used to assess overall functioning. The WHODAS 2.0 questionnaire comprises six domains with a five-point Likert-type scale (1 = no difficulty, 2 = mild, 3 = moderate, 4 = severe, and 5 = extreme) to measure the difficulty in performing activities. HIgher scores are associated with more disability.

SECONDARY OUTCOMES:
Sustainable change in substance use | 3 months, 6 months
  Assessed with the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool. TAPS consists of a combined screening component (TAPS-1) followed by a brief followed by a brief assessment (TAPS-2) for those who screen positive. Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance. TAPS Score Risk Category- 0=No Use in Past 3 Months, 1=Problem Use, 2+ =Higher Risk
Sustainable change in psychiatric symptom severity for a history of Major Depressive Disorder (MDD) | 3 months, 6 months
  The Patient Health Questionnaire (PHQ) will be used to assess this outcome. It is a multiple-choice self-report inventory that is used as a screening and diagnostic tool for mental health disorders of depression, anxiety, alcohol, eating, and somatoform disorders.There are 9 questions with a score from 0=Not al all to 3=Nearly everyday and one additional question about level of difficulty. Scores can range from 1 to 27 and are interpreted as: 1-4 Minimal depression, 5-9 Mild depression, 10-14 Moderate depression, 15-19 Moderately severe depression, and 20-27 Severe depression.
Sustainable change in psychiatric symptom severity given a history of bipolar disorder with the BDRS | 3 months, 6 months
  The Bipolar Depression Rating Scale (BPDS) has 20 questions with responses from 0= Nil to 3= Severe. The maximum score possible is 60. Higher scores indicate greater severity of symptoms.
Sustainable change in psychiatric symptom severity given a history of bipolar disorder with the YMRS | 3 months, 6 months
  The Young Mania Rating Scale (YMRS) has eleven items and is based on the patient's subjective report of his or her clinical condition, and generally limited to the previous 48 hours. Scores can range from 0 to 60 and higher scores are associated with more severe symptoms.
Sustainable change in psychiatric symptom severity for a history of post traumatic stress disorder (PTSD) | 3 months, 6 months
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) will be used to assess this outcome. The total severity score on the CAPS-5 represents the sum of the individual severity scores (0-4) for each of the 20 PTSD symptoms. Total scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Sustainable change in psychiatric symptom severity for a history of schizophrenia/schizophrenic disorders. | 3 months, 6 months
  The Positive and Negative Syndrome Scale (PANSS) will be used to asses this outcome. PANSS items are rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme); because the absence of symptoms is equal to 1 point, the lowest possible total score on both PANSS scales is 7. The range for both the negative and positive scales are 7 to 49.
Sustainable change in subjective quality of life | 3 months, 6 months
  The Quality of Life Scale (QOLS) will be used to assess this outcome. The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112. Higher score indicate higher quality of life.
Sustainable change in overall functioning | 3 months, 6 months
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) will be used to assess overall functioning. The WHODAS 2.0 questionnaire comprises six domains with a five-point Likert-type scale (1 = no difficulty, 2 = mild, 3 = moderate, 4 = severe, and 5 = extreme) to measure the difficulty in performing activities. HIgher scores are associated with more disability.
Feasibility of the drama therapy intervention | 12 weeks
  This outcome will be assessed by responses to an investigator developed structured interview with study staff at end of intervention.
Acceptability of the drama therapy intervention | 12 weeks
  This outcome will be assessed by responses to an investigator developed structured interview with study staff at end of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William-Bernard Reid-Varley, MD MPH, Principal Investigator — Boston Medical Center, Psychiatry Department
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No